CLINICAL TRIAL: NCT05512585
Title: A Physiological Study to Assess the Effects of Awake Prone Positioning in Healthy Volunteers Under Different Respiratory Support: A Randomized Crossover Study
Brief Title: A Physiological Study to Assess Awake Prone Positioning and Respiratory Support in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Jie Li, Associate Professor, Rush University Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APP-002
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: Prone positioning; high-flow nasal cannula; continuous positive airway pressure
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- awake prone positioning with room air (Active Comparator): Participants will stay in the prone position
  Interventions: Other: awake prone positioning with advanced respiratory support (high-flow nasal cannula or continuous positive airway pressure)
- awake prone positioning with high-flow nasal cannula (Experimental): Participants will stay in the prone position and breathe with high-flow nasal cannula
  Interventions: Other: awake prone positioning with advanced respiratory support (high-flow nasal cannula or continuous positive airway pressure)
- awake prone positioning with continuous positive airway pressure (Experimental): Participants will stay in the prone position and breathe with continuous positive airway pressure via face mask
  Interventions: Other: awake prone positioning with advanced respiratory support (high-flow nasal cannula or continuous positive airway pressure)
- supine position with room air (No Intervention): Participants will stay in the supine position
- supine position with high-flow nasal cannula (Active Comparator): Participants will stay in the supine position and breathe with high-flow nasal cannula
  Interventions: Other: awake prone positioning with advanced respiratory support (high-flow nasal cannula or continuous positive airway pressure)
- supine position with continuous positive airway pressure (Active Comparator): Participants will stay in the supine position and breathe with continuous positive airway pressure via face mask
  Interventions: Other: awake prone positioning with advanced respiratory support (high-flow nasal cannula or continuous positive airway pressure)

INTERVENTIONS:
Other: awake prone positioning with advanced respiratory support (high-flow nasal cannula or continuous positive airway pressure) — in this group, healthy subjects will stay in prone position for 20 mins with respiratory support of high-flow nasal cannula or CPAP
  Arms: awake prone positioning with continuous positive airway pressure; awake prone positioning with high-flow nasal cannula; awake prone positioning with room air; supine position with continuous positive airway pressure; supine position with high-flow nasal cannula

SUMMARY:
Awake prone positioning (APP) has been proven to reduce the intubation rate for patients with COVID-19-induced hypoxemic respiratory failure. Our recent meta-analysis found APP was only effective for patients who were treated by high-flow nasal cannula (HFNC), not for patients using conventional oxygen therapy (COT).In a recent multicenter RCT, Perkins and colleagues reported that continuous positive airway pressure (CPAP) was superior to HFNC and conventional oxygen therapy in reducing intubation rate. Thus, it is essential to evaluate the physiological mechanism of APP under different respiratory supports, such as COT, HFNC, or CPAP.

We hypothesize that HFNC or CPAP is more effective when combined with APP than COT combined with APP. Electrical impedance tomography (EIT imaging) has been broadly utilized to assess patient ventilation homogeneity and respiratory volume monitor (RVM) has been used to evaluate patient's tidal volumes breath-by-breath. In this study, 20 healthy volunteers will use different respiratory support devices (HFNC, CPAP, and COT) in different settings and their combinations withAPP in a random sequence, assessed by EIT and RVM.

DETAILED DESCRIPTION:
Awake prone positioning (APP) has been proven to reduce the intubation rate for patients with COVID-19-induced hypoxemic respiratory failure. Our recent meta-analysis found APP was only effective for patients who were treated by high-flow nasal cannula (HFNC), not for patients using conventional oxygen therapy (COT).In a recent multicenter RCT, Perkins and colleagues reported that continuous positive airway pressure (CPAP) was superior to HFNC and conventional oxygen therapy in reducing intubation rate. Thus, it is essential to evaluate the physiological mechanism of APP under different respiratory supports, such as COT, HFNC, or CPAP.

ELIGIBILITY:
Inclusion Criteria:

healthy adults aged between 21 to 65 years

Exclusion Criteria:

* Tested COVID positive within 21 days, or has any of the following symptoms in the last 21 days: sore throat, cough, chills, body aches for unknown reasons, shortness of breath for unknown reasons, loss of smell, loss of taste, fever at or greater than 100 degrees Fahrenheit.
* Currently have the following symptoms: sore throat, fever, coughing, shortness of breath, loss of smell or taste
* Non-English speaking
* Has any of the following diseases: asthma, chronic obstructive pulmonary disease, Uncontrolled Diabetes, hypertension, or untreated thyroid disease
* and spinal cord injury.
* Claustrophobia
* Pregnancy
* Pacemaker (EIT contraindication)
* face or chest skin injury that could not use a facemask or the electrode belt
* could not tolerate prone positioning for one hour

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
ventilation distribution assessed by EIT | 20 minutes
  Regional ventilation assessed by regional tidal impedance variations relative to global tidal impedance variation (ΔzROI/Δzglobal) obtained by electrical impedance tomography (EIT)

SECONDARY OUTCOMES:
tidal volume | 20 minutes
  the gas volume during tidal breathing
respiratory rates | 20 minutes
  breathing frequency during tidal breathing
comfort | 20 minutes
  subject's comfort which will be assessed by a 1-10 scale

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, PhD, Principal Investigator — Rush University
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perkins GD, Ji C, Connolly BA, Couper K, Lall R, Baillie JK, Bradley JM, Dark P, Dave C, De Soyza A, Dennis AV, Devrell A, Fairbairn S, Ghani H, Gorman EA, Green CA, Hart N, Hee SW, Kimbley Z, Madathil S, McGowan N, Messer B, Naisbitt J, Norman C, Parekh D, Parkin EM, Patel J, Regan SE, Ross C, Rostron AJ, Saim M, Simonds AK, Skilton E, Stallard N, Steiner M, Vancheeswaran R, Yeung J, McAuley DF; RECOVERY-RS Collaborators. Effect of Noninvasive Respiratory Strategies on Intubation or Mortality Among Patients With Acute Hypoxemic Respiratory Failure and COVID-19: The RECOVERY-RS Randomized Clinical Trial. JAMA. 2022 Feb 8;327(6):546-558. doi: 10.1001/jama.2022.0028. PMID 35072713
- [Background] Mauri T, Alban L, Turrini C, Cambiaghi B, Carlesso E, Taccone P, Bottino N, Lissoni A, Spadaro S, Volta CA, Gattinoni L, Pesenti A, Grasselli G. Optimum support by high-flow nasal cannula in acute hypoxemic respiratory failure: effects of increasing flow rates. Intensive Care Med. 2017 Oct;43(10):1453-1463. doi: 10.1007/s00134-017-4890-1. Epub 2017 Jul 31. PMID 28762180
- [Background] Riera J, Perez P, Cortes J, Roca O, Masclans JR, Rello J. Effect of high-flow nasal cannula and body position on end-expiratory lung volume: a cohort study using electrical impedance tomography. Respir Care. 2013 Apr;58(4):589-96. doi: 10.4187/respcare.02086. PMID 23050520
- [Background] Chiumello D, Chiodaroli E, Coppola S, Cappio Borlino S, Granata C, Pitimada M, Wendel Garcia PD. Awake prone position reduces work of breathing in patients with COVID-19 ARDS supported by CPAP. Ann Intensive Care. 2021 Dec 20;11(1):179. doi: 10.1186/s13613-021-00967-6. PMID 34928455
- [Background] Liu L, Xie J, Wang C, Zhao Z, Chong Y, Yuan X, Qiu H, Zhao M, Yang Y, Slutsky AS. Prone position improves lung ventilation-perfusion matching in non-intubated COVID-19 patients: a prospective physiologic study. Crit Care. 2022 Jun 29;26(1):193. doi: 10.1186/s13054-022-04069-y. No abstract available. PMID 35768877
- [Result] Ehrmann S, Li J, Ibarra-Estrada M, Perez Y, Pavlov I, McNicholas B, Roca O, Mirza S, Vines D, Garcia-Salcido R, Aguirre-Avalos G, Trump MW, Nay MA, Dellamonica J, Nseir S, Mogri I, Cosgrave D, Jayaraman D, Masclans JR, Laffey JG, Tavernier E; Awake Prone Positioning Meta-Trial Group. Awake prone positioning for COVID-19 acute hypoxaemic respiratory failure: a randomised, controlled, multinational, open-label meta-trial. Lancet Respir Med. 2021 Dec;9(12):1387-1395. doi: 10.1016/S2213-2600(21)00356-8. Epub 2021 Aug 20. PMID 34425070
- [Result] Li J, Luo J, Pavlov I, Perez Y, Tan W, Roca O, Tavernier E, Kharat A, McNicholas B, Ibarra-Estrada M, Vines DL, Bosch NA, Rampon G, Simpson SQ, Walkey AJ, Fralick M, Verma A, Razak F, Harris T, Laffey JG, Guerin C, Ehrmann S; Awake Prone Positioning Meta-Analysis Group. Awake prone positioning for non-intubated patients with COVID-19-related acute hypoxaemic respiratory failure: a systematic review and meta-analysis. Lancet Respir Med. 2022 Jun;10(6):573-583. doi: 10.1016/S2213-2600(22)00043-1. Epub 2022 Mar 16. PMID 35305308